CLINICAL TRIAL: NCT07340905
Title: Ethical Assessment Tool of Artificial Intelligence Impementation in Scientific Research
Brief Title: AI Ethical Assessment in Scientific Resreach
Acronym: AI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem ahmed, DR, Assiut University
Other Study IDs: AI
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Artificial Intelligence (AI)
Keywords: Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Artificial Intelligence (AI) is transforming scientific research by enabling computers to perform tasks that require human intelligence - such as data analysis, pattern recognition, prediction, and language processing.

AI is now integrated into every stage of the research process: from idea generation and literature review to data collection, analysis, and publication. Using tools like machine learning, deep learning, and natural language processing (NLP), researchers can analyze massive datasets, detect hidden trends, and accelerate discoveries across fields like medicine, biology, chemistry, and social sciences.

DETAILED DESCRIPTION:
The benefits of AI include speed, accuracy, efficiency, and innovation, allowing scientists to process information and generate hypotheses faster than ever. However, ethical challenges such as data bias, lack of transparency, accountability, plagiarism risks, and privacy concerns must be addressed through responsible AI governance.

ELIGIBILITY:
* Inclusion criteria
* Age ≥ 18
* Able to provide informed consent
* Has direct experience with research and/or AI tools used in research (often within the last 1-3 years)
* Speaks/reads the study language (e.g., English/Arabic)
* Available to complete the study activity (survey)
* Exclusion criteria
* No AI is involved.
* It's only theory/principles with no checklist or questions.
* It covers only one issue (privacy-only, bias-only) when you need full ethics.
* Not enough info to assess (no data source, no model description, no intended use).
* It's a small classroom/toy example with no real impact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Principal investigators / co-investigators
  Research assistants / lab members
  Data scientists / statisticians
  Students (Masters/PhD) working on AI-supported research
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Ethical Assessment Tool of Artificial Intelligence Impementation in Scientific Research | 6 months
  Ethical Assessment Tool of Artificial Intelligence Impementation in Scientific Research

REFERENCES:
- Available data/document: original article — https://pmc.ncbi.nlm.nih.gov/articles/PMC11370812/